



Participant Consent - Milk Intervention RCT

Thank you for agreeing to take part in this study. Please read the following consent form, initial wh

| nere ii | ndicated and sign if you are willing to participate. | , | |
|---|---|---|---|
| rategi | es to Improve Iodine Status in Early Pregnancy | Participant Number: | |
| | | Please | initial box |
| | I confirm that I have read, or had read to me, and understand th <a href="06.12.2021">06.12.2021</a> version 1.6 for the above study. I have had the oppo and have had these answered fully. | | |
| | I understand that my participation is voluntary, and I am free to without giving any reason and without my legal rights being affe | • | |
| | I understand the study is being conducted by researchers from Cand the Belfast Health and Social Care Trust, and that my persor securely on university premises and handled in accordance with 2018. | nal information will be held | |
| | I understand that data collected as part of this study may be loo individuals from Queen's University Belfast and regulatory authors to my taking part in this research. I give permission for these ind this information. | orities where it is relevant | |
| • | I agree to take part in the above study. | | |
| | I agree to my results being accessed using the clinical system 'La information being collected from the Northern Ireland Maternit | | |

06/12/2021 Version 1.4

## **CONFIDENTIAL**

| I agree to my GP being informed of my participation in the study and to my GP | | | study and to my GP being |
|---|---|---|---|
| informed of an | y abnormal te | st results. | |
| | | ation I provide may be publishe | · |
| publications. | wiii be maint | ained, and it will not be possibl | e to identify me from any |
| I understand th | I understand that this study is confidential but there are limits to confidentiality. Revelations | | |
| that are crimin<br>be broken by t | | | may require confidentiality to |
| I agree to gift r | d I consent to the storage and | | |
| use of my sample for future research. I understand that I will not benefit financially from any research. If you do not want your samples to be stored for future research, you can still participate in the current study. | | | |
| <ul> <li>I agree to being contacted later and invited to take part in future studies of a similar nature</li> <li>I understand that I am only agreeing to receive information and I am under no obligation</li> </ul> | | | |
| to take part in | any future stu | dies, if you decide not to conse | ent to being contacted in the |
| Name of Participant (p | lease print) | Signature | Date |
| Name of Person taking consent | | Signature | Date |
| (please print) | | | |
| Chief Investigator: | Professor Jay | yne Woodside | |
| | j.woodside@ | qub.ac.uk | |

Version 1.4 06/12/2021